CLINICAL TRIAL: NCT02590133
Title: A Multi-institutional, Randomized Controlled, Phase II Clinical Trial on Comparison of Efficacy and Safety of Nedaplatin Plus 5-Fu Combined With and Without Endostar® Continuous Intravenous Infusion in Refractory Nasopharyngeal Carcinoma
Brief Title: A Phase II Clinical Trial of Chemotherapy With or Without Endostar® Continuous Intravenous Infusion in Refractory NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yun-fei Xia (Other)
Responsible Party: Sponsor-Investigator, Yun-fei Xia, Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2015-031-01
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Refractory Nasopharyngeal Carcinoma, Endostar, 5-Fu
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endostatins; endostar protein; Fluorouracil; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nedaplatin+5-Fu+Endostar (Experimental): Drug: Recombinant Human Endostatin Injection (Endostar) Endostar, 15mg/m2/d, continuous intravenous infusion in 2ml/h for 30 days each cycle, 60 days as one cycle, 6 cycles in total Drug: Fluorouracil (5-Fu) 5-Fu, 200mg/m2/d, continuous intravenous infusion in 2ml/h for 30 days each cycle, 60 days as one cycle, 6 cycles in total Drug: Nedaplatin Nedaplatin, 80mg/m2/d, intravenous drip on d1 and d28 each cycle, 60 days as one cycle, 6 cycles in total
  Interventions: Drug: Recombinant Human Endostatin Injection (Endostar); Drug: Fluorouracil (5-Fu); Drug: Nedaplatin
- Nedaplatin+5-Fu (Active Comparator): Drug: Fluorouracil (5-Fu) 5-Fu, 200mg/m2/d, continuous intravenous infusion in 2ml/h for 30 days each cycle, 60 days as one cycle, 6 cycles in total Drug: Nedaplatin Nedaplatin, 80mg/m2/d, intravenous drip on d1 and d28 each cycle, 60 days as one cycle, 6 cycles in total
  Interventions: Drug: Fluorouracil (5-Fu); Drug: Nedaplatin

INTERVENTIONS:
Drug: Recombinant Human Endostatin Injection (Endostar) — 15mg/m2/d, continuous intravenous infusion in 2ml/h for 30 days each cycle, 60 days as one cycle, 6 cycles in total
  Other Names: Endostar
  Arms: Nedaplatin+5-Fu+Endostar
Drug: Fluorouracil (5-Fu) — 200mg/m2/d, continuous intravenous infusion in 2ml/h for 30 days each cycle, 60 days as one cycle, 6 cycles in total
  Other Names: 5-Fu
Drug: Nedaplatin — 80mg/m2/d, intravenous drip on d1 and d28 each cycle, 60 days as one cycle, 6 cycles in total
  Other Names: Nedaplait

SUMMARY:
We define refractory nasopharyngeal carcinoma as the following: recurrence with radiation brain injury after radiotherapy, recurrence after the second or more courses of radiotherapy, standard treatment failure after recurrence, and first-line treatment failure after multiple distant metastasis.

There is no standard treatment for refractory nasopharyngeal carcinoma. Platinum plus 5-Fu is the classic regimen for primary treatment of nasopharyngeal carcinoma.

Endostatin is a multiple targeted angiogenesis inhibitor acting on tumor associated neovascular endothelial cells, normalizing the morphology and function of tumor vasculature, and indirectly leading to the quiescence or reduction of tumors.

The purpose of this phase II clinical trial is to determine the efficacy and safety of nedaplatin plus continuous low dose 5-Fu intravenous infusion combined with endostar® (Recombinant Human Endostatin Injection) continuous intravenous infusion compared with nedaplatin plus continuous low dose 5-Fu intravenous infusion alone in refractory nasopharyngeal carcinoma.

The study hypothesis is that nedaplatin plus continuous low dose 5-Fu intravenous infusion combined with endostar® continuous intravenous infusion is effective and safe in refractory nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
With the extension of survival time in nasopharyngeal carcinoma(NPC), more and more patients suffer from recurrence with radiation brain injury after radiotherapy, recurrence after the second or more courses of radiotherapy, standard treatment failure after recurrence, and first-line treatment failure after multiple distant metastasis. We define these four types as refractory nasopharyngeal carcinoma[1-2] due to the complex and high risk of treatment and poor prognosis. For recurrence and metastasis NPC, the objective response rate ranges from 25% to 46.4% with platinum-based, or 5-Fu-based, or gemcitabine-based salvage chemotherapy[2--5].

At present, there is no standard treatment for refractory nasopharyngeal carcinoma.

Most patients in this trial were pretreated with cisplatin-based chemotherapy. Nedaplatin has the equivalent antitumor effect with cisplatin and less renal toxicity and gastrointestinal toxicity in the treatment of NPC[6]. In addition, nedaplatin does not have the cross tolerance with cisplatin. After cisplatin failure, nedaplatin(80-100 mg/m2) still work in NPC treatment[3].

5-Fu is a classic, effective, and safe chemotherapeutic drug in NPC treatment. Low dose continuous intravenous infusion of 5-Fu(300mg/m2/d, 6 weeks) is a effective regimen for recurrent and metastasis NPC with low toxicity[4].

Endostatin is a multiple targeted angiogenesis inhibitor acting on tumor associated neovascular endothelial cells, normalizing the morphology and function of tumor vasculature, and indirectly leading to the quiescence or reduction of tumors[7-9]. Anti-angiogenic therapy might optimally require that endothelial cells be exposed to steady blood levels of the inhibitor, and blood levels of certain angiogenesis inhibitors (such as endostatin) that are too high or too low will be ineffective[7,10]. Endostar® is recombinant human endostatin injection with better medicinal properties, stability and curative effect. Hoekman K. etc conducted a phase I clinical pharmacokinetic study in advanced cancer and the results showed that continuous intravenous pump of endostar® is safe[11]. Moreover, endostar® combined with chemotherapy can improve the outcome of the chemotherapy alone and does not increase the treatment related toxicity, such as in advanced non-small-cell lung cancer[12], advanced cervical cancer[13], advanced gastric cancer[14] and also metastasis NPC[15].

Given that the patients in this trial have the following features: had received standard radical treatment, poor tolerance of treatment due to the toxicity after many courses of chemotherapy, and the present treatment goal is palliative therapy. Therefore, the treatment principle in this trial is using low toxicity, well tolerance treatment regimen to relieve and control tumor, improve the quality of life, and further to prolong the survival time.

Based on above background and considering the Efficacy and tolerability, we use nedaplatin plus continuous low dose 5-Fu intravenous infusion as chemotherapy regimen, and administrate endostar® in continuous intravenous infusion.

This phase II randomized controlled trial is to investigate the efficacy and safety of nedaplatin plus continuous low dose 5-Fu intravenous infusion combined with endostar® (Recombinant Human Endostatin Injection) continuous intravenous infusion compared with nedaplatin plus continuous low dose 5-Fu intravenous infusion alone in refractory nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients have provided a signed Informed Consent Form.
* Histologically confirmed diagnosis of refractory nasopharyngeal carcinoma (the best), or when histology is difficult to obtained, the following clinical diagnosis of refractory nasopharyngeal carcinoma must be confirmed: clear and directional clinical symptoms, at least two kinds of imaging diagnosis on the basis of magnetic resonance (MR), and clear and directional signs.
* Age: 18-70 years old.
* Without dysfunction of heart, lung, liver, kidney, and hematopoiesis, and normal electrocardiogram.
* Karnofsky Performance Scores ≥ 50, Life expectancy ≥ 3 months, tolerance to at least two cycles of chemotherapy.
* At least one measurable tumor based on RECIST 1.1 ( longest diameter: ≥20 mm by CT or magnetic resonance (MR) scan)
* No history of serious allergic to biologic agents
* No history of other malignant tumors, except cured cervical carcinoma in situ and basal skin cancer.

Exclusion Criteria:

* Having the serious cardiovascular disease or other serious complications.
* Woman in pregnancy and breast-feeding.
* Allergic to intervention drugs and dextran.
* Patients participated in clinical trials of other drugs within 4 weeks.
* Use of other chemotherapy drugs, biological treatment, and Chinese medicine anti-cancer drugs at the same time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
objective response (OR) rate based on Recist 1.1 edition | From the date of first drug administration, evaluation of response was performed every cycle during the treatment and then every 3 months after the completion of the treatment up to 36 months
  include complete remission and partial remission

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | From the date of first drug administration, evaluation of response was performed every cycle during the treatment and then every 3 months after the completion of the treatment up to 36 months
  include complete remission, partial remission, and progressive disease
Progress Free Survival (PFS) | From the date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  3 years PFS
Overall Survival (OS) | From the date of first drug administration until the date of death, assessed up to 36 months
  3 years OS
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From the date of first drug administration, evaluation was performed every cycle during the treatment and then every 3 months after the completion of the treatment up to 36 months, using NCI CTCAE version 4.0
  Safety evaluation according to NCI Common Terminology Criteria (CTC) 4.0
Quality of life | From the date of first drug administration, evaluation was performed every cycle during the treatment and then every 3 months after the completion of the treatment up to 36 months, using EORTC quality of life questionnaire (QLQ)-C30
  Quality of life evaluation according to EORTC quality of life questionnaire (QLQ)-C30

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, Prof, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang F, Wu K, Gao F, Zhang W, Shi F, Li C. Refractory nasopharyngeal carcinoma: positron emission tomography combined with computed tomography-guided 125I seed implantation therapy after repeated traditional radiochemotherapy. Otolaryngol Head Neck Surg. 2013 Sep;149(3):417-23. doi: 10.1177/0194599813491221. Epub 2013 May 28. PMID 23715683
- [Background] Gao Y, Huang HQ, Bai B, Cai QC, Wang XX, Cai QQ. Treatment outcome of docetaxel, capecitabine and cisplatin regimen for patients with refractory and relapsed nasopharyngeal carcinoma who failed previous platinum-based chemotherapy. Expert Opin Pharmacother. 2014 Feb;15(2):163-71. doi: 10.1517/14656566.2014.866652. Epub 2013 Dec 3. PMID 24295173
- [Background] Peng PJ, Ou XQ, Chen ZB, Liao H, Peng YL, Wang SY, Zhang HY, Lin Z. Multicenter phase II study of capecitabine combined with nedaplatin for recurrent and metastatic nasopharyngeal carcinoma patients after failure of cisplatin-based chemotherapy. Cancer Chemother Pharmacol. 2013 Aug;72(2):323-8. doi: 10.1007/s00280-013-2203-0. Epub 2013 Jun 1. PMID 23728706
- [Background] Fandi A, Taamma A, Azli N, Bachouchi M, Yanes B, Armand JP, Cvitkovic E. Palliative treatment with low-dose continuous infusion 5-fluorouracil in recurrent and/or metastatic undifferentiated nasopharyngeal carcinoma type. Head Neck. 1997 Jan;19(1):41-7. doi: 10.1002/(sici)1097-0347(199701)19:13.0.co;2-v. PMID 9030944
- [Background] Chen C, Wang FH, Wang ZQ, An X, Luo HY, Zhang L, Chen YC, Xu RH, Li YH. Salvage gemcitabine-vinorelbine chemotherapy in patients with metastatic nasopharyngeal carcinoma pretreated with platinum-based chemotherapy. Oral Oncol. 2012 Nov;48(11):1146-51. doi: 10.1016/j.oraloncology.2012.05.021. Epub 2012 Jun 27. PMID 22748450
- [Background] Zheng J, Wang G, Yang GY, Wang D, Luo X, Chen C, Zhang Z, Li Q, Xu W, Li Z, Wang D. Induction chemotherapy with nedaplatin with 5-FU followed by intensity-modulated radiotherapy concurrent with chemotherapy for locoregionally advanced nasopharyngeal carcinoma. Jpn J Clin Oncol. 2010 May;40(5):425-31. doi: 10.1093/jjco/hyp183. Epub 2010 Jan 19. PMID 20085903
- [Background] Folkman J. Angiogenesis: an organizing principle for drug discovery? Nat Rev Drug Discov. 2007 Apr;6(4):273-86. doi: 10.1038/nrd2115. PMID 17396134
- [Background] Folkman J. Antiangiogenesis in cancer therapy--endostatin and its mechanisms of action. Exp Cell Res. 2006 Mar 10;312(5):594-607. doi: 10.1016/j.yexcr.2005.11.015. Epub 2005 Dec 22. PMID 16376330
- [Background] Peng F, Xu Z, Wang J, Chen Y, Li Q, Zuo Y, Chen J, Hu X, Zhou Q, Wang Y, Ma H, Bao Y, Chen M. Recombinant human endostatin normalizes tumor vasculature and enhances radiation response in xenografted human nasopharyngeal carcinoma models. PLoS One. 2012;7(4):e34646. doi: 10.1371/journal.pone.0034646. Epub 2012 Apr 9. PMID 22496834
- [Background] Kisker O, Becker CM, Prox D, Fannon M, D'Amato R, Flynn E, Fogler WE, Sim BK, Allred EN, Pirie-Shepherd SR, Folkman J. Continuous administration of endostatin by intraperitoneally implanted osmotic pump improves the efficacy and potency of therapy in a mouse xenograft tumor model. Cancer Res. 2001 Oct 15;61(20):7669-74. PMID 11606410
- [Background] Hansma AH, Broxterman HJ, van der Horst I, Yuana Y, Boven E, Giaccone G, Pinedo HM, Hoekman K. Recombinant human endostatin administered as a 28-day continuous intravenous infusion, followed by daily subcutaneous injections: a phase I and pharmacokinetic study in patients with advanced cancer. Ann Oncol. 2005 Oct;16(10):1695-701. doi: 10.1093/annonc/mdi318. Epub 2005 Jul 12. PMID 16012180
- [Background] Rong B, Yang S, Li W, Zhang W, Ming Z. Systematic review and meta-analysis of Endostar (rh-endostatin) combined with chemotherapy versus chemotherapy alone for treating advanced non-small cell lung cancer. World J Surg Oncol. 2012 Aug 24;10:170. doi: 10.1186/1477-7819-10-170. PMID 22917490
- [Background] Ke QH, Zhou SQ, Huang M, Lei Y, Du W, Yang JY. Early efficacy of Endostar combined with chemoradiotherapy for advanced cervical cancers. Asian Pac J Cancer Prev. 2012;13(3):923-6. doi: 10.7314/apjcp.2012.13.3.923. PMID 22631672
- [Background] Xu R, Ma N, Wang F, Ma L, Chen R, Chen R, Kebinu M, Ma L, Han Z, Ayixiamu, Mayier M, Su P, Naman Y, Jieensi H, Yang H, Adili A, Aili S, Liu J. Results of a randomized and controlled clinical trial evaluating the efficacy and safety of combination therapy with Endostar and S-1 combined with oxaliplatin in advanced gastric cancer. Onco Targets Ther. 2013 Jul 25;6:925-9. doi: 10.2147/OTT.S46487. Print 2013. PMID 23926435
- [Background] Jin T, Li B, Chen XZ. A phase II trial of Endostar combined with gemcitabine and cisplatin chemotherapy in patients with metastatic nasopharyngeal carcinoma (NCT01612286). Oncol Res. 2013;21(6):317-23. doi: 10.3727/096504014X13983417587401. PMID 25198661